CLINICAL TRIAL: NCT04008901
Title: A Single-center, Randomized, Double-blind, Placebo-controlled, Intervention Study for the Efficacy and Safety of "BST104" (Lonicera Flos Extract) in Mild to Moderate Functional Dyspepsia Subjects
Brief Title: The Efficacy and Safety of "BST104" (Lonicera Flos Extract) in Mild to Moderate Functional Dyspepsia Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BST104-01
Record Dates: First submitted 2019-06-02; First posted 2019-07-05 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Functional Dyspepsia; Irritable Bowel Syndrome
Keywords: Functional dyspepsia; Irritable Bowel Syndrome; Lonicera Flos; GSRS; Antioxidant
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: This study is a single center, random assignment, double blind placebo human application study. If a subject agrees in writing to participate in the human aptitude test, the medical examination required in accordance with the human aptitude test plan were conducted and randomly assigned only to those who are suitable for the selection criteria. The randomly assigned target was given a Lonicera Flos extract (BST104) 250 mg/day or placebo for eight weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Random assignment, double blind placebo human application study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Active Comparator): The randomly assigned target was given a Lonicera Flos extract (BST104) 175 mg/day for eight weeks.
  Interventions: Drug: BST-104 (Lonicera Flos Extract)
- Placebo group (Placebo Comparator): The randomly assigned target was given a placebo for eight weeks.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: BST-104 (Lonicera Flos Extract) — 175 mg of Lonicera Flos extract in 1 tablet (300 mg)
  Arms: Treatment group
Drug: Placebo oral tablet — 0 mg of Lonicera Flos extract in 1 tablet (300 mg)
  Arms: Placebo group

SUMMARY:
This study was conducted to prove the efficacy of BST-104 in patients with mild to moderate FD.

DETAILED DESCRIPTION:
In this single center, double-blind, randomized clinical trial, patients diagnosed with FD using Rome III criteria were allocated to either test group (300 mg of BST-104, containing 175 mg of Flos Lonicera extracts, twice daily) or placebo group (300 mg placebo, twice daily). Male and female patients > 19 years of age who had mild to moderate FD were eligible. They had baseline endoscopic screening, and patients without active lesions (peptic ulcer disease or gastric erosions) were enrolled. Written informed consent was obtained from all participants.

ELIGIBILITY:
Inclusion Criteria:

* Persons who was diagnosed with functional indigestion in adult over 19 years of age and did not require early medication was conducted with the participation

Exclusion Criteria:

* Persons who is allergic to natural substances and substances
* Persons who need treatment for reflux esophagitis, gastric ulcer, and acute gastritis according to gastroscopy findings
* Persons with past history of stomach or esophagus surgery, or patients who are unable to take esophagogastroduodenoscopy
* Persons who continue to apply medications that can cause ulcers such as steroids, nonsteroidal anti-inflammatory drugs and aspirin (Patients taking low-dose aspirin for prevention of cardiovascular disease were allowed)
* Persons diagnosed with malignant tumors within five years
* Persons who drink more than four times a week
* Severe liver failure (more than 2 .5 times the normal upper limit of ALT, AST, γGT)
* In case of a severe renal failure, including chronic or acute kidney failure
* Persons with uncontrolled diabetes, cerebrovascular disease,
* Persons diagnosed with diseases requiring surgery within three months
* Zollinger Ellison sy n drome, esophageal stenosis, duodenal ulcer, pancreatitis, absorption disorder, or malignant disease in the gastrointestinal tract
* Pregnant women, nursing mothers, having plans for pregnancy
* In case of participating another human study within four weeks

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-11-08 (Actual)

PRIMARY OUTCOMES:
GSRS total score improvement : GSRS score at baseline - GSRS score after 8 weeks of administration | 8 weeks
  GSRS (Gastrointestinal Symptom Rating Scale) total score improvement after 8 weeks of administration, compared to Baseline
  GSRS is consisted of 15 upper and lower gastrointestinal symptoms, and each item is rated on a 7-point Likert scale, 0 = no symptoms, 7 = worst
  Total score scale : 0~105 (15x7), 0 = no symptoms, 105 = worst, decreased score is considered as improvement, increased score is considered as worsening
  stomach pain (0~7) heartburn (0~7) acid reflux (0~7) hunger pain (0~7) nausea (0~7) rumbling (0~7) bloating (0~7) burping (0~7) flatus (0~7) constipation (0~7) diarrhea (0~7) loose stools (0~7) hard stools (0~7) urgency (need to have a bowel movement) (0~7) sensation of not completely emptying the bowels (0~7)
  total score (sum of 15 symptoms scores, 0~105)

SECONDARY OUTCOMES:
GSRS improvement rate : (total GSRS score at baseline - total GSRS score after 8 weeks of administration) / GSRS score at baseline | 8 weeks
  Total GSRS score improvement rate after 8 weeks of administration, compared to Baseline
Improvement of 15 individual symptom scores of GSRS : symptom score at baseline - symptom score after 8 weeks | 8 weeks
  15 individual symptoms of upper and lower abdominal discomfort after 8 weeks of administration, compared to Baseline
Changes in serum antioxidant and anti-inflammatory marker level | 8 weeks
  Changes in serum antioxidant (8-OHdG, Thiobarbituric acid reactive substances (TBARS), total antioxidant, hs-CRP level) after 8 weeks of administration, compared to baseline
Changes in dyepepsia-related quality of life | 8 weeks
  Changes in dyepepsia-related quality of life using NDI (Nepean Dyspepsia Index) questionnaire after 8 weeks of administration, compared to baseline
  NDI-K (Nepean Dyspepsia Index Korean) is consisted of 5 categories and 25 questions of gastrointestinal symptoms, with each question is rated on a 5-point Likert scale, 0 = worst, 5 = no symptoms
  Total score scale : (sum of individual question score) x 100/125
  0~100, 0 = worst condition, 100 = no symptoms, decreased score is considered as worsening, increased score is considered as improvement
  Interference daily activities/work (0~30) Knowledge/control (0~20) Eating/drinking (0~15) Sleep disturbance (0~45) Work/study (0~15)
  Total score (sum of individual question score) x 100/125

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Choi Y, Kim N, Noh GT, Lee JY, Lee DH. The Efficacy and Safety of GCWB104 (Flos Lonicera Extract) in Functional Dyspepsia: A Single-Center, Randomized, Double-Blind, Placebo-Controlled Study. Gut Liver. 2020 Jan 15;14(1):67-78. doi: 10.5009/gnl19283. PMID 31945816